CLINICAL TRIAL: NCT04364217
Title: Evaluating the Mechanism of Pain and Itch Reduction in Burn Scars Following Fractional Ablative CO2 Laser Treatment
Brief Title: Pain and Itch Reduction in Burn Scars Treated With Fractional CO2 Laser
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in enrollment lead to withdrawing the study without enrollment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Friedstat, Instructor of Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019P003424
Record Dates: First submitted 2020-03-06; First posted 2020-04-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hypertrophic Scar; Burn Scar
Keywords: Pain; Itch
MeSH Terms: conditions — Cicatrix, Hypertrophic; Pain; Pruritus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Other): Laser treatment to 3x3cm2 area. It will receive the Luminous ultra pulse fractional ablative carbon dioxide laser at 150mJ, 3% density and 250Hz
  Interventions: Device: Luminis ultrapulse fractional ablative carbon dioxide laser

INTERVENTIONS:
Device: Luminis ultrapulse fractional ablative carbon dioxide laser — This laser will target water molecules and ablate columns of tissue that are approximately 3mm deep.
  Other Names: Fractional CO2 laser treatment

SUMMARY:
Hypertrophic Burn Scars (HTBS) are often treated with Fractional CO2 laser therapy to improve cosmetic appearance. It has been noted that this leads to a reduction in the pain and itch associated with this type of scars. While this phenomenon is commonly described in the literature, the mechanism of pain and itch reduction in unclear. The investigators aim to better understand this process by histological evaluation of HTBS at different stages of laser treatment.

DETAILED DESCRIPTION:
During our study, patients with painful and/or itchy burn scars will undergo standard treatment with fractional CO2 laser. In addition to the standard of care treatment, participants will undergo skin biopsies and be asked to complete Patient Reported Outcome Measure questionnaires related to their HTBS. Burn scars will also undergo standard and 3 dimensional photography at the different stages of treatment. Biopsy samples will undergo various staining techniques to establish the changes in tissue that occur with the laser treatment. This information will also be correlated with the symptomatic changes.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a hypertrophic burn scar treated by skin grafts or allowed to heal secondarily
* Burn must have occurred within the last 2 years from time of recruitment
* Patient must have symptoms of pain and/or itch and/or hypersensitivity in the hypertrophic burn scar area
* Patient must already be planning to undergo laser treatment for their burn scar
* Patient must be willing to undergo biopsy procedures
* Patient must be willing and able to participate in the study with a year of follow-up
* Not be pregnant or planning to become pregnant during the treatment phase of the study

Exclusion Criteria:

* Medical Conditions that preclude laser treatment
* Active tanning, including the use of tanning booths, during the course of the study
* Inability to complete surveys
* Previous laser (PDL, CO2), surgical reconstructive treatment procedures done on the hypertrophic burn scar
* Current treatment with other procedures or drugs (experimental or other) in area of interest
* Medications that interfere with wound healing (oral steroids, immunosuppressive medications, chemotherapy or other)
* Medication for itch (steroids, antihistamines, or other)
* Medication for pain (opioids, topical pain treatment, gabapentin, ondasetron, paroxetine or other)
* Adverse reactions to topical or local anesthetic agents needed for this study, if no alternative to the said agent exists
* The study area should not be part of a contracture or other hypertrophic scar that would be better treated with surgical procedures.
* The study scar must not be adjacent to/in continuity with areas of HTBS that are planning to be treated with surgical interventions.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject
* Patient suffers from epilepsy or seizure disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Histological change in nerve density | 7 months
  The investigators will stain the collected skin with markers specific to nerves to in order to count the number of nerves per biopsy area.
Histological change in nerve morphology | 7 months
  The investigators will stain the collected skin with markers specific to nerves to in order to compare the size and shape of cutaneous nerves before and after treatment. This will be based on subjective evaluation and not a predetermined scale.

SECONDARY OUTCOMES:
Symptomatic Improvement Assessment | 7 months
  Patient Reported Outcome Measures will be collected via the Patient and Observer Scar Assessment Scale (POSAS). This is a validated questionnaire that includes 5 physician-completed parameters and 6 patient-reported measures. Each parameter is rated from 1-10 with a score of 1 representing "skin that appears close to normal" and 10 representing the "worst scare imaginable". Overall, the final score will range from 11( best outcome) to 110 (worst outcome).
  Physician parameters relate to the scar appearance such as color and thickness of the scar; while the patient-reported parameters also include symptomatic factors, such as degree of pain associated with the scar

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Friedstat, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States